CLINICAL TRIAL: NCT02377999
Title: Safety and Efficacy of Repeat Use of Picato® 0.05% in the Treatment of Anogenital Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXP-1167
Record Dates: First submitted 2015-02-20; First posted 2015-03-04 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Anogenital Warts
MeSH Terms: conditions — Condylomata Acuminata | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment of genetial warts with Picato (Experimental)
  Interventions: Drug: Picato

INTERVENTIONS:
Drug: Picato

SUMMARY:
An exploratory open label, single treatment trial of anogenital warts with Picato® repeated up to 2 times with two weeks intervals.

DETAILED DESCRIPTION:
The purpose of the present trial is to explore the safety, tolerability and efficacy when treating GW with Picato® 0.05% gel. The primary outcome measures will be related to safety and tolerability and consists of severity of any local reactions in the treated area; treatment-related adverse events (AEs) and serious AEs.

ELIGIBILITY:
Inclusion Criteria:

* 1. A clinical diagnosis of external anogenital/perianal warts with at least 2 warts and no more than 20 warts located in one or more of the following anatomic locations:

  1. In both sexes: inguinal, perineal, and perianal areas
  2. In men: penis shaft, scrotum, glans penis and foreskin
  3. In women: on the vulva
* 2. Subjects has a total wart areas of at least 10 mm2, but not more than 500 mm2
* 3. Female subjects of childbearing potential must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment

Exclusion Criteria:

* 1. Subject has received any topical and/or destructive treatments for external anogenital warts within 4 weeks (within 12 months for imiquimod and within 12 weeks for sinecatechins) prior to enrolment
* 2. Subject suffer from any of the following conditions:

  1. Known human immunodeficiency virus (HIV) infection
  2. An outbreak of herpes genitalis in the wart areas within 4 weeks prior to enrolment
  3. Has internal (rectal urethral, vaginal/cervical) warts that require or are undergoing treatment
  4. Has a dermatological disease (e.g. psoriasis) or skin condition in the wart areas
* 3. Subjects using systemic virostatic compounds or immunosuppressive medication within 30 days prior to enrollment
* 4. Prior quadrivalent HPV vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of incidence and severity of Local Skin Reactions (LSR) | Measured two weeks after every treatment and final measurement 2 weeks after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, Professor MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en